CLINICAL TRIAL: NCT01059695
Title: Retrospective Analysis of Treatment and Quality of Life of Women Treated for Cervical Carcinoma FIGO Stage IB-1 to IVb From 2000-2008 in Limburg, a Province in the South of the Netherlands.
Brief Title: Analysis of the Results of Treatment for Cervical Carcinoma in Limburg
Acronym: CervixLimburg
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); Atrium Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-24-09/12
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; retrospective; quality of life; treatment
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Analysis of all women treated for cervical cancer between 2000 and 2008 in Limburg, a province in the south of the Netherlands. Patient characteristics, diagnosis, treatment modalities, complications and survival will be analyzed by record review. Quality of life of the living study population will be assessed using the EORTC QLQ-C30 and QOQ-CX24 questionnaire. Patients will be identified via registration data from the Integraal Kankercentrum Limburg.

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer FIGO stage IB-1 to IVB
* Treated in Limburg between 2000 and 2008

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women diagnosed with cervical cancer FIGO stage IB-1 to IV between 2000 and 2008 in Limburg, a province in the south of the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Quality of life
  Quality of life of the living study population will be assessed using the EORTC QLQ-C30 and QOQ-CX24 questionnaire